CLINICAL TRIAL: NCT04969198
Title: UW Withdraw From Tobacco Study: Enhancing and Evaluating Tobacco Withdrawal Assessment Psychometrics and Validity
Brief Title: UW Withdraw From Tobacco Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-0792; A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison); 5R01HL109031 (NIH); Protocol Version 2/21/2022 (Other: UW Madison)
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2023-11

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotine Patch + Nicotine Mini Lozenge (Experimental): No medication for 1 Week after Target Quit Day (TQD). Medication started 1 Week after TQD.
  Patches (Nicotine): 14 mg Patches for 4 weeks postquit (Week 1-5), then 7 mg patches for 4 weeks (Week 6-9)
  Mini Lozenge (Nicotine): 2 mg Mini Lozenges 5x per day (up to 20x day max) for 8 weeks post quit (Week 1-9)
  Interventions: Drug: Combination nicotine replacement therapy (Nicotine patch + nicotine mini-lozenge)

INTERVENTIONS:
Drug: Combination nicotine replacement therapy (Nicotine patch + nicotine mini-lozenge) — Nicotine patch and mini-lozenge dosing will be based off the 2008 Public Health Services (PHS) Clinical Practice Guideline and package insert with adjustments to account for the delayed start 1-week post-TQD. All participants will receive 2mg mini-lozenge due to the superior palatability of the 2mg lozenges. Participants are encouraged to use at least 5 mini-lozenges per day for the full 8 weeks. Participants who report any smoking or nicotine use (e.g., even a cigarette puff, e-cigarette use) in the 3 days before C-NRT distribution will receive 4 weeks of 14mg and 4 weeks of 7mg nicotine patches. Participants who report complete abstinence from smoking and nicotine in the 3 days before C-NRT distribution will receive 8 weeks of 7mg nicotine patches.
  Other Names: C-NRT

SUMMARY:
It is of considerable scientific and clinical importance to assess tobacco withdrawal accurately since withdrawal severity is highly determinant of smoking cessation success. In addition, smoking cessation pharmacotherapy produces its effects on smoking abstinence by suppressing such symptoms. However, in order to ensure that a measure of tobacco withdrawal is sensitive to severe withdrawal, it is essential to examine a period of unmedicated abstinence. The current study aims to validate, and possibly enhance, a revised Wisconsin Smoking Withdrawal Scale long and brief version for use in research and clinical settings.

Two hundred adults who smoke cigarettes daily and report a desire to quit smoking will be enrolled. This is a treatment-delay, one-group clinical trial that is intended to enhance the assessment of tobacco withdrawal amongst participants who try to quit smoking with delayed use of cessation medication. Participants will not receive any pharmacotherapy during the first 1 week of their quit attempt and will initiate 8 weeks of combination nicotine replacement therapy (C-NRT; nicotine patch + nicotine mini-lozenge) starting 1 week past the target quit day (TQD). Participants will receive 4 counseling sessions as well (1 pre-quit, 3 post-quit). Participants will complete 4 weeks of ecological momentary assessment (EMA) smartphone surveys including a 2-week baseline (starting TQD-14) and 2-week post-TQD (1-week un-medicated, 1-week using C-NRT).

ELIGIBILITY:
Inclusion Criteria:

* Smoke ≥5 cigarettes per day for past year
* ≥21 years old
* Able to read and write English
* Desire to quit smoking
* Not currently engaged in cessation treatment
* Eligible to use combination nicotine replacement therapy
* Willing and able to attend study visits
* Have reliable smartphone access
* Not currently pregnant, trying to get pregnant, or breastfeeding
* Willing to respond to ecological momentary assessment prompts and other study activities
* Baseline breath carbon monoxide (CO) ≥5ppm

Exclusion Criteria:

* Used pipe tobacco, cigars, snuff, or chew more than twice in the past week
* Used e-cigarette, vaping, or any other electronic nicotine delivery product more than twice in the past week
* Unwilling to try to abstain from all non-medicinal nicotine use (including e-cigarettes) for the duration of the Cessation Phase (other than nicotine replacement therapy provided by the study)
* Currently taking varenicline or bupropion
* Allergy to adhesive tape
* Previous reaction to the nicotine patch or mini-lozenge that prevented them from continuing to use it
* Unwilling to use study approved methods of birth control while taking study medication and for 1 month after discontinuing study medication [only for women of child-bearing potential]
* Hospitalized for a stroke, heart attack, congestive heart failure, ulcers, or diabetes within the last year
* History of seizure within the last year
* Diagnosis of and/or treatment for schizophrenia, other psychotic disorders, or bipolar disorder within the last 5 years
* End-stage renal disease
* Suicide attempt or suicidal ideation within the last 12 months
* Severe hypertension > 180/100 mmHg

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Baker, PhD, Principal Investigator — University of Wisconsin, Madison; Jesse T Kaye, PhD, Study Director — University of Wisconsin, Madison
Locations (1):
- Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will preregister their study design and publish the study protocol along with the publication of the primary outcome paper. Finally, investigators will make de-identified data and analysis code publicly available on the Open Science Framework (OSF: https://osf.io) or similar platform in accordance with NIH policy and principles of transparent science practices

REFERENCES:
- See also: University of Wisconsin Center for Tobacco Research and Intervention — https://ctri.wisc.edu/researchers/studies/withdraw-from-tobacco-study/

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Patch + Nicotine Mini Lozenge: No medication for 1 Week after Target Quit Day (TQD). Medication started 1 Week after TQD.
  Patches (Nicotine): 14 mg Patches for 4 weeks postquit (Week 1-5), then 7 mg patches for 4 weeks (Week 6-9)
  Mini Lozenge (Nicotine): 2 mg Mini Lozenges 5x per day (up to 20x day max) for 8 weeks post quit (Week 1-9)
  Combination nicotine replacement therapy (Nicotine patch + nicotine mini-lozenge): Nicotine patch and mini-lozenge dosing will be based off the 2008 Public Health Services (PHS) Clinical Practice Guideline and package insert with adjustments to account for the delayed start 1-week post-TQD. All participants will receive 2mg mini-lozenge due to the superior palatability of the 2mg lozenges. Participants are encouraged to use at least 5 mini-lozenges per day for the full 8 weeks. Participants who report any smoking or nicotine use (e.g., even a cigarette puff, e-cigarette use) in the 3 days before C-NRT distribution will receive 4 weeks of 14mg and 4 weeks of 7mg nicotine patches. Participants who report complete abstinence from smoking and nicotine in the 3 days before C-NRT distribution will receive 8 weeks of 7mg nicotine patches.
Period: Overall Study
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Started | 232
Number Participants for 2 Weeks Pre-quit Timepoint Analysis | 218
Number Participants for 1 Week Pre-quit Timepoint Analysis | 208
Number Participants for 1-3 Days Pre-quit Timepoint Analysis | 199
Number Participants for 1-2 Days Post-quit Timepoint Analysis | 198
Number Participants for 1 Week Post-quit Timepoint Analysis | 195
Number Participants for 2 Weeks Post-quit Timepoint Analysis | 186
Number Participants for 9 Weeks Post-quit Timepoint Analysis | 176
Completed | 176
Not Completed | 56
Not completed — Withdrawal by Subject | 20
Not completed — Withdrawn by PI for Participant Non-Compliance | 16
Not completed — Lost to Follow-up | 20

BASELINE CHARACTERISTICS:
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 184
  >=65 years | 48
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 116
  Female | 112
  Other | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 221
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 187
  More than one race | 6
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Score on Wisconsin Smoking Withdrawal Scale2 Long (WSWS2-L)
Description: Self-reported withdrawal symptom severity in the last 24 hours using the Wisconsin Smoking Withdrawal Scale 2(WSWS-2) Long Version.
  WSWS-2 consists of 19 items. Each item answers on a scale from 1=not at all to 7=extremely, how much a participant has been bothered in the last 24 hours. Mean score from 1-7 is reported. Higher scores indicate more severe withdrawal symptoms.
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 2.64 (1.13)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 2.36 (1.02)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 2.29 (1.03)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.69 (1.57)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.73 (1.29)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 2.32 (1.05)

2. Primary Outcome: Change in Wisconsin Smoking Withdrawal Scale2 Brief Score
Description: Self-reported withdrawal symptom severity in the last 24 hours using the Wisconsin Smoking Withdrawal Scale 2(WSWS-2) Brief Version.
  WSWS-2 consists of 6 items. Each item answers on a scale from 1=not at all to 7=extremely, how much a participant has been bothered in the last 24 hours. Higher scores indicate more severe withdrawal symptoms.
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 2.69 (1.27)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 2.38 (1.15)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 2.33 (1.15)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.74 (1.25)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.72 (1.21)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 2.29 (1.08)

3. Secondary Outcome: Change in WSWS2-L Subscale Score : Craving
Description: Self-reported withdrawal symptom severity subscales (negative affect, craving, hunger, sleep, restlessness, concentration) in the last 24 hours using the Wisconsin Smoking Withdrawal Scale 2 Long Version. Each item answers on a scale from 1=not at all to 7=extremely, how much a participant has been bothered in the last 24 hours.
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 4.55 (1.75)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 4.12 (1.75)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 3.98 (1.75)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 4.86 (1.76)
  1 week post-quit: number analyzed (Participants) | 193
  1 week post-quit | 4.47 (1.8)
  2 weeks post-quit: number analyzed (Participants) | 184
  2 weeks post-quit | 3.3 (1.69)

4. Secondary Outcome: Change in WSWS2-L Subscale Score : Negative Affect
Description: as for outcome 3
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 2.13 (1.41)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 1.95 (1.33)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 1.92 (1.21)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.35 (1.48)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.48 (1.6)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 2.06 (1.26)

5. Secondary Outcome: Change in WSWS2-L Subscale Score : Concentration
Description: as for outcome 3
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 1.94 (1.28)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 1.73 (1.11)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 1.74 (1.28)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.04 (1.43)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.18 (1.56)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 1.86 (1.17)

6. Secondary Outcome: Change in WSWS2-L Subscale Score : Sleep Problems
Description: as for outcome 3
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 2.73 (1.63)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 2.35 (1.44)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 2.24 (1.47)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.37 (1.49)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.55 (1.58)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 2.37 (1.4)

7. Secondary Outcome: Change in WSWS2-L Subscale Score: Hunger
Description: as for outcome 3
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 2.39 (1.46)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 2.19 (1.38)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 2.06 (1.23)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.34 (1.4)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.44 (1.42)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 2.39 (1.39)

8. Secondary Outcome: Change in WSWS2-L Subscale Score : Restlessness
Description: as for outcome 3
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 2.13 (1.41)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 1.95 (1.33)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 1.92 (1.21)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 2.35 (1.48)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.48 (1.6)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 2.06 (1.26)

9. Secondary Outcome: 9-Week Point-Prevalence Abstinence: Number of Participants Who Were Abstinent
Description: Biochemically confirmed self-reported total abstinence from any cigarette use (even a single puff) for the seven days preceding the target follow up day, confirmed with carbon monoxide reading of less than or equal to 5 ppm.
Time Frame: 9 weeks after quit date
Population: Investigators use 'intent-to-treat' analysis for this outcome measure so people who are lost to follow up are counted as still smoking (not abstinent).
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
Participants | 46

10. Secondary Outcome: Change in Total Score on Minnesota Tobacco Withdrawal Scale (MTWS)
Description: Self-reported withdrawal symptom severity in the last 24 hours using the Minnesota Tobacco Withdrawal Scale (MTWS). MTWS consists of 17 items. Mean score from 0 to 4 is reported. Higher scores indicate more severe withdrawal symptoms.
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 216
  2 weeks pre-quit | 0.965 (0.89)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 0.855 (0.83)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 0.837 (0.83)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 1.16 (0.93)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 1.2 (0.95)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 1.00 (0.84)

11. Secondary Outcome: Change in WSWS2-L Subscale Score: Anhedonia
Description: Exploratory subscale of the WSWS2-L, self-reported withdrawal symptom severity subscales (negative affect, craving, hunger, sleep, restlessness, concentration) in the last 24 hours using the Wisconsin Smoking Withdrawal Scale 2 Long Version. Each item answers on a scale from 1=not at all to 7=extremely, how much a participant has been bothered in the last 24 hours.
Time Frame: pre-quit (2 weeks, 1 week, 1-3 days) and post-quit (1-2 days, 1 week, 2 weeks)
Population: Not all participants contributed data for each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
Number analyzed (Participants) | 232
score on a scale
  2 weeks pre-quit: number analyzed (Participants) | 217
  2 weeks pre-quit | 1.93 (1.46)
  1 week pre-quit: number analyzed (Participants) | 208
  1 week pre-quit | 1.75 (1.41)
  1-3 days pre-quit: number analyzed (Participants) | 199
  1-3 days pre-quit | 1.65 (1.37)
  1-2 days post-quit: number analyzed (Participants) | 198
  1-2 days post-quit | 1.91 (1.5)
  1 week post-quit: number analyzed (Participants) | 195
  1 week post-quit | 2.03 (1.49)
  2 weeks post-quit: number analyzed (Participants) | 185
  2 weeks post-quit | 1.79 (1.22)

ADVERSE EVENTS:
Time Frame: All participants were assessed for adverse events at all study visits over the course of 10 weeks.
Arm/Group | Nicotine Patch + Nicotine Mini Lozenge
All-Cause Mortality (participants affected / at risk) | 0/232
Serious Adverse Events (participants affected / at risk) | 8/232
Other Adverse Events (participants affected / at risk) | 96/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch + Nicotine Mini Lozenge (N=232)
Kidney Stones (Renal and urinary disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Campylobacter Colitis (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation and heart failure (Cardiac disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch + Nicotine Mini Lozenge (N=232)
Nausea (Gastrointestinal disorders) | 24 (24)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 10 (10)
Headache (General disorders) | 11 (14)
Weakness (General disorders) | 8 (8)
Heartburn (Gastrointestinal disorders) | 4 (4)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Coughing (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Hiccup (General disorders) | 5 (5)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gas (Gastrointestinal disorders) | 1 (1)
Rapid, Slow, Pounding or Irregular Heartbeat (Cardiac disorders) | 2 (2)
Itching or Hives (Skin and subcutaneous tissue disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 1 (1)
Swelling or tingling in mouth or throat (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Chest Tightness (General disorders) | 2 (2)
Trouble Breathing (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Skin Rash, Irritation, or Swelling (Skin and subcutaneous tissue disorders) | 7 (7)
Insomnia/Distrupted Sleep/Vivid Dreams (Nervous system disorders) | 33 (38)
Changes in Mood/Agitation or Distress (General disorders) | 17 (17)
Suicidal Ideation (General disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT04969198/Prot_001.pdf
  • Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT04969198/SAP_000.pdf
  • Informed Consent Form (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT04969198/ICF_002.pdf